CLINICAL TRIAL: NCT07010276
Title: Centromedian Deep Brain Stimulation vs. Vagus Nerve Stimulation for the Treatment of Drug-Resistant Epilepsy and Epileptic Spasms in Children: A Randomized Trial
Brief Title: Deep Brain Stimulation vs. Vagus Nerve Stimulation for Epileptic Spasms
Acronym: DBS-VNS-ES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, George Ibrahim, Staff Neurosurgeon, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000080101
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy; Seizure
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VNS Treatment (Active Comparator): Patients in the VNS treatment arm will undergo surgical VNS implantation.
  Interventions: Device: VNS arm
- DBS Treatment (Active Comparator): Patients in the DBS treatment arm will undergo surgical DBS implantation.
  Interventions: Device: DBS Arm

INTERVENTIONS:
Device: DBS Arm — Patients in the DBS treatment arm will undergo surgical DBS implantation.
  Arms: DBS Treatment
Device: VNS arm — Patients in the VNS treatment arm will undergo surgical VNS implantation.
  Arms: VNS Treatment

SUMMARY:
Deep Brain Stimulation vs. Vagus Nerve Stimulation for the Treatment of Drug-Resistant Epilepsy and Epileptic Spasms in Children: A Randomized Control Trial

DETAILED DESCRIPTION:
To directly compare the effectiveness and safety of deep brain stimulation (DBS) vs. vagus nerve stimulation (VNS) in children with drug-resistant epilepsy (DRE) or epileptic spasms.

This will be an open, non-blinded randomized control trial. Twenty (20) patients will be recruited and enrolled in this pilot study from SickKids.

Expected study duration is 36-48 months.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male patients 5 years of age and over (17 and 11 months), not including 18 years old
* Diagnosis of drug-resistant epilepsy with failure after trial of two anti-epileptic
* Medications (as defined by Kwan et al. 20093). All children screened for entry into the study will be re-diagnosed by a neurologist prior to entry.
* Main seizure type includes epileptic spasms and tonic spasms, as confirmed by electroencephalography.
* Parents or legal guardians, including caregivers, are informed and able to give written consent.
* Ability to comply with all testing, follow-ups and study appointments and protocols for 12 months following the end of the duration of the study

Exclusion Criteria:

* Substance dependence or abuse in the last 6 months, excluding caffeine and nicotine
* Any contraindication to MRI scanning. A preoperative MRI scan is essential to
* Planning DBS and therefore any contraindication to MRI is a contraindication to enrollment in the study.
* Unwillingness or inability to return to SickKids for follow-up visits.
* Presence of cardiac arrhythmias, or other cardiac, respiratory, renal or endocrine conditions that will result in significant risk from a surgical procedure.
* Pregnancy
* Inability to communicate adequately in English in order to complete the baseline and follow-up questionnaires.
* A co-morbid condition that requires frequent MRI scanning as part of the patient's regular care.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
McHugh Scale for outcome measure after Vagal Nerve Stimulation | 1 year
  The McHugh Scale is a system used by doctors to assess how much a patient's seizures have improved after receiving Vagal Nerve Stimulation (VNS) therapy. Similar to the Engel Scale for epilepsy surgery, it categorizes outcomes into different classes based on the percentage reduction in seizure frequency, helping to standardize the evaluation of VNS treatment effectiveness.
Engel Epilepsy Surgery Outcome Scale | 1 year
  The Engel Epilepsy Surgery Outcome Scale is a common way doctors classify how well epilepsy surgery worked for a patient. It uses different classes (I, II, III, IV) to describe the reduction in seizures after surgery, ranging from being completely seizure-free to having no worthwhile improvement.
  Class I: Seizure-free Class II: Rare seizures Class III: Significant improvement but not seizure-free Class IV: No improvement or worse
ILAE Classification | 1 year
  he ILAE Classification is a standardized system used by doctors worldwide to precisely describe and categorize seizures and epilepsy. It helps them understand where a seizure starts in the brain, if a person's awareness is affected, and what symptoms occur, which then guides the best treatment plan.
Quality of Life in Childhood Epilepsy Questionnaire (QOLCE) | 1 year
  The QOLCE is designed to evaluate the health-related quality of life specifically in children with epilepsy, covering various aspects impacted by their condition.

SECONDARY OUTCOMES:
Hague Seizure Severity Scale (HASS) - parent-perception scale | 1 year
  The HASS is a patient-reported outcome measure used to quantify the overall severity of epileptic seizures, considering aspects like seizure type, frequency, and impact.
Seizure Severity Questionnaire (SSQ) | 1 year
  The SSQ is a self-report questionnaire that assesses the severity of epileptic seizures based on the patient's perception of their seizures and their impact on daily life.
Pediatric Quality of Life Inventory (PedsQL) | 1 year
  A parent questionnaire designed to evaluate health-related quality of life in children.
  Scores range from 0 to 92, with higher scores indicating poorer quality of life.
CarerQoL - measure of caregiver quality of life | 1 year
  This instrument measures the subjective well-being and quality of life experienced by informal caregivers, focusing on both the positive and negative impacts of their caregiving role.
The Child Health Utility 9D (CHU9D) | 1 year
  The Child Health Utility 9D (CHU9D) is a survey for kids and teens (ages 7-17) that asks simple questions about their health and how they feel. This helps us understand their overall "quality of life" and allows researchers to compare the benefits of different treatments by measuring "Quality-Adjusted Life Years" (QALYs), which is like getting a score for how healthy and long a life someone lives.

CONTACTS AND LOCATIONS:
Overall Officials: George M Ibrahim, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada